CLINICAL TRIAL: NCT04560998
Title: Effects of Semaglutide on Functional Capacity in Patients With Type 2 Diabetes and Peripheral Arterial Disease
Brief Title: A Research Study to Compare a Medicine Called Semaglutide Against Placebo in People With Peripheral Arterial Disease and Type 2 Diabetes
Acronym: STRIDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9535-4533; 2019-003399-38 (Registry Identifier: European Medicines Agency (EudraCT)); U1111-1238-7071 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-09-18; First posted 2020-09-23 (Actual); Results first posted 2025-07-08 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2; Peripheral Arterial Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Peripheral Arterial Disease | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): Semaglutide given in addition to standard-of-care treatment
  Interventions: Drug: Semaglutide
- Placebo (semaglutide) (Placebo Comparator): Placebo given in addition to standard-of-care treatment
  Interventions: Drug: Placebo (semaglutide)

INTERVENTIONS:
Drug: Semaglutide — Semaglutide is administered subcutaneously (s.c.; under the skin) once-weekly for 52 weeks in a dose escalating manner: 0.25 mg from week 1 to week 4, 0.5 mg from week 5 to week 8 and 1.0 mg from week 9 to week 52.
  Arms: Semaglutide
Drug: Placebo (semaglutide) — Placebo (semaglutide) is administered s.c. once-weekly for 52 weeks in a dose escalating manner: 0.25 mg from week 1 to week 4, 0.5 mg from week 5 to week 8 and 1.0 mg from week 9 to week 52.
  Arms: Placebo (semaglutide)

SUMMARY:
This study is done to see if semaglutide has an effect on walking ability compared with placebo (dummy medicine) in people with peripheral arterial disease (PAD) and type 2 diabetes. Participants will either get semaglutide or placebo ("dummy") medicine - which treatment participants get is decided by chance. Semaglutide is a medicine for type 2 diabetes that can be prescribed by doctors in some countries. Participants will get the study medicine (semaglutide or placebo) in a pre-filled pen for injection. Participants must inject it once a week into the stomach area, thigh, or upper arm, at any time of the day. The study will last for about 59 weeks. Participants will have 8 clinic visits and 1 phone call with the study doctor. At some clinic visits, participants will have blood tests. At some visits participants will also do a treadmill test to measure how far they can walk. Women cannot take part if pregnant, breast-feeding or planning to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age above or equal to 18 years at the time of signing informed consent. For Japan: Male or female, age above or equal to 20 years at time of signing informed consent
* Diagnosed with type 2 diabetes mellitus at least 180 days prior to the day of screening.
* Symptomatic PAD with intermittent claudication corresponding to Fontaine stage IIa (Rutherford classification grade I, category 1 and 2) meeting all of the following:

  1. Stable symptoms of PAD with intermittent claudication in Fontaine stage IIa (able to walk without stopping more than 200 m/656 feet/2 blocks) for at least 90 days prior to the day of screening based on patient interview.
  2. Screening flat treadmill test (3.2 km/h (2 mph)): Pain-free walking distance of at least 200 meters/656 feet.
  3. Screening constant load treadmill test with fixed inclination of 12% and a fixed speed of 3.2 km/h (2 mph): Walking distance equal to or less than 600 meters/1968 feet.
  4. Ankle-brachial-index (ABI) equal to or below 0.90 or toe-brachial index (TBI) equal to or below 0.7 (the leg with lowest index is chosen in case of bilateral disease).

Exclusion Criteria:

* Current or previous treatment with any GLP-1 receptor agonist (GLP-1-RA) within 90 days prior to the day of screening.
* Walking ability limited by conditions other than PAD (e.g. aortic aneurism, dysregulated arrhythmia or hypertension, angina pectoris, heart failure, chronic obstructive or restrictive pulmonary disease, Parkinson's disease, severe peripheral neuropathy, amputations, wheel chair or walker dependency, osteoarthritis, morbid obesity, severe varicose veins, etc.).
* Planned orthopaedic surgery in the legs, or other major surgery known on the day of screening (surgery affecting walking ability).
* Vascular revascularisation procedure of any kind 180 days prior to the day of screening.
* Planned arterial revascularisation known on the day of screening.
* Myocardial infarction, stroke, hospitalisation for unstable angina pectoris or transient ischemic attack within 180 days prior to the day of screening.
* Heart failure presently classified as being in New York Heart Association (NYHA) class III-IV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 792 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (1452), Study Director — Novo Nordisk A/S
Locations (194):
- United States (43):
  - Cardiology, PC, Birmingham, Alabama
  - Central Arkansas Veteran's Healthcare System, Little Rock, Arkansas
  - Cardio Innovation & Resch Ctr, Long Beach, California
  - Angel City Research, Inc., Los Angeles, California
  - St. Joseph Heritage Healthcare_Mission Viejo, Mission Viejo, California
  - Rocky Mount Reg VA Med-DN, Aurora, Colorado
  - Univ of Colorado at Denver, Aurora, Colorado
  - Bay Area Cardiology Associates, P.A., Brandon, Florida
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Tampa Bay Medical Research, Clearwater, Florida
  - Jacksonville Ctr For Clin Res, Jacksonville, Florida
  - DMI Research, Pinellas Park, Florida
  - University of South Florida, Tampa, Florida
  - Accel Research Site-Georgia, Eatonton, Georgia
  - Reg Infectious Dis Infuse Ctr, La Grange, Georgia
  - Aiyan Diabetes Center, Martinez, Georgia
  - Endeavor Health Glenbook Hosp, Glenview, Illinois
  - Central IL Diabetes and Clinical Research, Springfield, Illinois
  - Cardiovascular Rsrch of NW_IN, Munster, Indiana
  - Central Cardio Assoc HPS, Elizabethtown, Kentucky
  - Cambridge Medical Trials, Alexandria, Louisiana
  - LOUISIANA HEART Center, Covington, Louisiana
  - Clinical Trials of Ame, LLC, Monroe, Louisiana
  - Ascension Saint Agnes Heart Ca, Baltimore, Maryland
  - Boston Medical Center_Cary, Boston, Massachusetts
  - Minneapolis Cardiology Assoc, Minneapolis, Minnesota
  - Amicis Centers of Clinical Research, St Louis, Missouri
  - Nebraska West Iowa Hlth System, Omaha, Nebraska
  - Methodist Phys Clin Heart Cons, Omaha, Nebraska
  - Dartmouth-Hitchcock Med Ctr, Lebanon, New Hampshire
  - NYU Langone Med Assoc Chelsea, New York, New York
  - Accellacare_NC, Wilmington, North Carolina
  - Capital Area Research LLC, Camp Hill, Pennsylvania
  - Penn Presb Med Ctr, Philadelphia, Pennsylvania
  - Vanderbilt U Med Ctr_Nashville, Nashville, Tennessee
  - PharmaTex Research, Amarillo, Texas
  - Northwest Houston Cardiology, P.A., Houston, Texas
  - Houston Heart & Vascular Associates, Humble, Texas
  - Texas Cardiology Associates of Houston, Kingwood, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - North Dallas Research Associates, McKinney, Texas
  - Victoria Heart and Vasc Ctr, Victoria, Texas
  - Selma Medical Associates, Winchester, Virginia
- Austria (4):
  - Universitätsklinik für Innere Medizin Graz, Graz
  - Univ.-Klinik für Innere Medizin III, Innsbruck
  - Klinik Landstraße, Vienna
  - AKH Wien, Vienna
- Belgium (6):
  - Imeldaziekenhuis Bonheiden - Thoracic and Vascular Surgery, Bonheiden
  - Ziekenhuis Oost-Limburg AV - Thoracic, Genk
  - UZ Gent - Thoracale Vasculaire Heelkunde, Ghent
  - UZ Gent_Gent_1, Ghent
  - AZ Groeninge - Thoracic Vascular Surgery, Kortrijk
  - UZ Leuven - Hart en Vaatziekten, Leuven
- Canada (10):
  - North York Diagn & Cardiac Ctr, North York, Ontario
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - The Ottawa Hospital, Civic Campus, Ottawa, Ontario
  - ViaCar Recherche Clinique Inc, Brossard, Quebec
  - Ecogene-21, Chicoutimi, Quebec
  - Clinique Sante Cardio MC, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - CISSS des Laurentides, Saint-Jérôme, Quebec
  - CHU de Quebec-Universite Laval, Québec
  - Institut universitaire de cardiologie, Québec
- China (7):
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - The First Bethune hospital of Jilin University-Endocrinology, Changchun, Jilin
  - The first hospital of Jilin University, Changchun, Jilin
  - 1st Affiliated Hosp of Xi'an JiaoTong Uni Medical College, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an JiaoTong University-Cardiovascular, Xi'an, Shaanxi
  - Tianjin Union Medical Center-Cardiology, Tianjin
  - Tianjin Union Medicine Centre, Tianjin
- Czechia (5):
  - CTC Hodonin s.r.o., Hodonín
  - EDUMED Jaromer, Jaroměř
  - Kucera, Ostrava Dubina
  - Diabetologicka ambulance Plzen, Pilsen
  - II. interni klinika - klinika kardiologie a angiologie 1. LF, Prague
- Denmark (4):
  - Kolding Sygehus Karkirurgi, Kolding
  - Rigshospitalet Karkirurgisk afd. RK 3111, København Ø
  - Hjerte-, Lunge- og Karkirurgisk afdeling T, Odense
  - Regionshospitalet Viborg - Karkirurgisk Afsnit, Viborg
- Germany (10):
  - Kardiologische Praxis, Bad Homburg
  - Herz- und Diabeteszentrum NRW - Bad Oeynhausen, Bad Oeynhausen
  - Kreutzmann, Dresden
  - Uniklinik TU Dresden - Med. Klinik und Poliklinik III Angiologie, Dresden
  - MVZ CCB Frankfurt und Main-Taunus GbR, Frankfurt
  - Uniklinik Schleswig-Holstein - Medizinischen Klinik I am Campus Lübeck, Lübeck
  - Universitätsmedizin der JGU Mainz - Kardiologie I, Mainz
  - Institut für Diabetesforschung GmbH Münster - Dr. med. Rose, Münster
  - Gemeinschaftspraxis Haggenmiller/Jeserich, Nuremberg
  - Zentrum für klinische Studien Alexander Segner, Saint Ingbert-Oberwürzbach
- Greece (8):
  - University Hospital of Athens ATTIKON, Athens, Attica
  - "Laiko" General Hospital of Athens, Athens
  - Konstantopouleio G.H. of Athens, "Agia Olga", Athens
  - "Hygeia" General Hospital of Athens, Athens
  - General Hospital of Chios "Skilitsio" - Cardiology Clinic, Chios
  - General Hospital of Lamia, Lamia
  - 'Ippokrateio' General Hospital of Thessaloniki, Thessaloniki
  - General Hospital of Thessaloniki "G.Papanikolaou", Thessaloniki
- Hungary (6):
  - Szegedi Tudományegyetem II. sz Belgyógyászati és Kardiológia, Szeged, Csongrád-Csanád
  - Léda Platán Magánklinika, Zalaegerszeg, Zala County
  - Szent Margit Rendelőintézet Nonprofit Kft., Budapest
  - Szent Imre Egyetemi Oktatókórház Angiológia, Budapest
  - Semmelweis Egyetem Városmajori Szív- és Érgyógyászat, Budapest
  - Coromed SMO Kft., Pécs
- India (11):
  - Sanjeevani Superspeciality Hospital, Ahmedabad, Gujarat
  - Shri B D Mehta Mahavir Heart Institute, Surat, Gujarat
  - Shri B. D. Mehta Mahavir Heart Institute, Surat, Gujarat
  - Shri Krishna Hrudayalaya & Critical Care Centre, Nagpur, Maharashtra
  - Shrikrishna Hrudayalaya and critical care centre, Nagpur, Maharashtra
  - Vijan Hospital & Research Centre, Nashik, Maharashtra
  - VMMC & Safdarjung Hospital, New Dehli, New Delhi
  - SP Medical College, Bikaner, Rajasthan
  - Osmania General Hospital, Hyderabad, Telangana
  - Udyaan Health Care, Lucknow, Uttar Pradesh
  - Sir Ganga Ram Hospital, New Delhi
- Japan (14):
  - New Tokyo Heart Clinic_Matsudo-shi, Chiba,, Chiba
  - Akaicho Clinic, Chiba-shi, Chiba
  - Takahashi Hospital_Cardiology, Hyōgo
  - Higashi Takarazuka Satoh Hospital_Cardiology, Hyōgo
  - Higashi Takarazuka Satoh Hospital, Hyōgo
  - Naka Kinen Clinic_Internal medicine, Ibaraki
  - Naka Kinen Clinic, Ibaraki
  - Nishiyamado Keiwa Hospital_Internal Medicine, Ibaraki
  - Omihachiman Community Medical Center_Omihachiman-shi, Siga, Omihachiman-shi, Siga
  - Minamiosaka Hospital_Internal medicine, Osaka
  - Saitama Cardiovascular and Respiratory Center, Saitama
  - Omi Medical Center_Cardiovascular Medicine, Shiga
  - Omi Medical Center, Shiga
  - Minamino Cardiovascular Hospital_Cardiovascular medicine, Tokyo
- Stradini PAD, Riga, Latvia
- Malaysia (7):
  - Hospital Universiti Sains Malaysia, Kota Bharu, Kelantan
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - University Technology MARA (UiTM) - Sg Buloh, Sungai Buloh, Selangor
  - National Heart Institute, Kuala Lumpur
  - Hospital Queen Elizabeth II, Sabak Bernam
- Norway (3):
  - Haukeland universitetssykehus - Karkirurgisk avdeling, Bergen
  - Sørlandet sykehus HF Kristiansand, Kristiansand
  - OUS, Aker, Oslo
- Poland (8):
  - Med. Cent. Diabet. Endo. Metabol. DIAB-ENDO-MET, Krakow, Lesser Poland Voivodeship
  - UniCardia & UniMedica & UniEstetica, Krakow
  - Centrum Medyczne OMEDICA, Poznan
  - Velocity Nova Sp. z o.o., Puławy
  - Gabinety Lekarskie LabMed, Szczecin
  - Narodowy Instytut Kardiologii Stefana kardynała Wyszynskiego, Warsaw
  - DoktorA, Warsaw
  - Centrum Badan Klinicznych, Wroclaw
- Russia (21):
  - Multispecialty Medical Clinic Anturium LLC, Barnaul
  - Road Clinical Hospital at station Chelyabinsk, Chelyabinsk
  - Irkutsk State Medical Academy of Postgraduate Education, Irkutsk
  - Limited Liability Company "Alliance Biomedical Ural Group", Izhevsk
  - SRMC "Your Health" LLC, Kazan'
  - FSBI 'I.I. Dedov National Medical Research Center of Endocrinology' of the MH of Russia, Moscow
  - Federal Bureau for Medical and Social Expertise, Moscow
  - Pirogov Russian National Research Medical University MoH, Moscow
  - LLC RC Medical, Novosibirsk
  - SGIoH of Novosibirsk region "CC Hospital #19", Novosibirsk
  - State Novosibirsk regional clinical hospital, Novosibirsk
  - LLC "Clinical diagnostic center Ultramed", Omsk
  - Ryazan State Medical University, Ryazan
  - Joint Stock Company "Polyclinic Complex", Saint Petersburg
  - Limited Liability Company "Clinic" MEDINEF ", Saint Petersburg
  - Limited Liability Company "Energiya Zdoroviya", Saint Petersburg
  - SGHI "Polyclinic #106", Saint Petersburg
  - Regional clinical cardiology dispensary, Saratov
  - SHI Saratov City Clinical Hospital #9, Saratov
  - Voronezh Regional Clinical Consultive-diagnostic Centre, Voronezh
  - Polyclinic #2 in Yoshkar-Ola, Yoshkar-Ola
- Spain (7):
  - Centro Periférico de Especialidades Bola Azul, Almería
  - Hospital Reina Sofia, Córdoba
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Civil de Málaga, Málaga
  - Hospital Virgen de la Macarena, Seville
  - Hospital Vithas Sevilla, Seville
- Sweden (2):
  - Kärlkirurgen/kärllab, Gothenburg
  - Kärlmottagningen, Uppsala
- Taiwan (7):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Kuang Tien General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital_main, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou Branch, Taoyuan District
- Thailand (10):
  - Srinagarind Hospital, Muang, Changwat Khon Kaen
  - King Chulalongkorn Memorial Hospital, Cardiology department, Bangkok
  - Phramongkutklao Hospital-cardio, Bangkok
  - Research Institute for Health Sciences, CMU, Chiang Mai
  - Rihes - Research Institute for Health Sciences, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
  - Maharat Nakhon Ratchasima Hospital_Ratchasima, Nakhon Ratchasima
  - Maharat Nakhon Ratchasima Hospital_, Nakhon Ratchasima
  - Thammasat University Hospital_Pathumthani, Pathum Thani
  - Songklanagarind Hospital, Songkhla

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Bonaca MP, Catarig AM, Houlind K, Ludvik B, Nordanstig J, Ramesh CK, Rasouli N, Sourij H, Videmark A, Verma S; STRIDE Trial Investigators. Semaglutide and walking capacity in people with symptomatic peripheral artery disease and type 2 diabetes (STRIDE): a phase 3b, double-blind, randomised, placebo-controlled trial. Lancet. 2025 May 3;405(10489):1580-1593. doi: 10.1016/S0140-6736(25)00509-4. Epub 2025 Mar 29. PMID 40169145

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 129 sites in 21 countries.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive treatment with either semaglutide or placebo as an adjunct to standard-of-care.
Groups:
- Semaglutide: Participants received once-weekly (OW) subcutaneous injection (s. c.) of semaglutide for 52 weeks. Participants received a dose of 0.25 milligrams (mg) from week 0 to week 4, then the dose was increased to 0.5 mg from week 4 to week 8. From week 8 to week 52, the dosage was 1.0 mg.
- Placebo: Participants received once-weekly (OW) subcutaneous injection (s. c.) of placebo matched for semaglutide for 52 weeks.
Period: Overall Study
Arm/Group | Semaglutide | Placebo
Started | 396 | 396
Full Analysis Set (FAS included all randomised participants. All participants were analyzed according to the treatment to which they were assigned at randomisation.) | 396 | 396
Safety Analysis Set | 396 | 395
Completed (Participants attended follow-up visit or died during trial considered completers in the trial.) | 366 | 379
Not Completed | 30 | 17
Not completed — Withdrawal by Subject | 18 | 12
Not completed — Lost to Follow-up | 8 | 5
Not completed — Physician Decision | 4 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomised participants. All participants were analyzed according to the treatment to which they were assigned at randomisation
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide | Placebo | Total
Number analyzed (Participants) | 396 | 396 | 792
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.2 (9.71) | 67.0 (8.96) | 66.6 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 88 | 195
  Male | 289 | 308 | 597
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 388 | 385 | 773
  Unknown or Not Reported | 1 | 5 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 131 | 109 | 240
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 4 | 8
  White | 259 | 279 | 538
  Other | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximum Walking Distance on a Constant Load Treadmill Test
Description: Change in maximum walking distance on a constant load treadmill test is presented. The constant-load treadmill test with fixed speed (3.2 km/h, 2 mph) and fixed inclination (12%) is a standardised method for functional assessment of patients with peripheral artery disease. Participants continue on the treadmill after indicating onset of pain and should continue as long as possible until pain limits further activity. This distance is noted as the maximum walking distance. The outcome measure was evaluated based on data from in-study observation period. In-study observation period is defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: Baseline (week 0), end of treatment (week 52)
Population: Full Analysis Set (FAS). Overall Number of Participants Analyzed = number of participants with available data for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Ratio of maximum walking distance
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 338 | 345
Ratio of maximum walking distance | 1.21 [0.95 to 1.55] | 1.08 [0.86 to 1.36]
Statistical Analysis 1: Comparison: Semaglutide vs Placebo; Test type: Superiority; p = 0.0004, Wilcoxon (Mann-Whitney); The Hodges-Lehmann estimate = 1.13, 95% CI 2-sided [1.056 to 1.211]

2. Secondary Outcome: Follow-up Change in Maximum Walking Distance on a Constant Load Treadmill Test
Description: Change in maximum walking distance on a constant load treadmill test is presented. The constant-load treadmill test with fixed speed (3.2 km/h, 2 mph) and fixed inclination (12%) is a standardised method for functional assessment of patients with peripheral artery disease. Participants continue on the treadmill after indicating onset of pain and should continue as long as possible until pain limits further activity. This distance is noted as the maximum walking distance. The outcome measure was evaluated based on data from in-study observation period. In-study observation period is defined as the period from date of randomisation to one of the following dates, which-ever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: Baseline (week 0), end of follow-up (week 57)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Ratio of maximum walking distance
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 329 | 333
Ratio of maximum walking distance | 1.16 [0.92 to 1.48] | 1.10 [0.87 to 1.40]
Statistical Analysis 1: Comparison: Semaglutide vs Placebo; Test type: Superiority; p = 0.0380, Wilcoxon (Mann-Whitney); The Hodges-Lehmann estimate = 1.08, 95% CI 2-sided [1.004 to 1.156]

3. Secondary Outcome: Change in Vascular Quality of Life Questionnaire-6 (VascuQoL-6) Score
Description: Change in VascuQoL-6 score is presented. VascuQoL-6 is a peripheral artery disease-specific questionnaire with 6 items covering social, emotional, functional as well as pain- and symptom-related aspects of the patient´s overall quality of life. Each item has a 4-point response scale (where 1 = worst score and 4 = best score). The endpoint analysed is the total score (range: 6-24) generated by summing the scores from all items. A higher score indicates better health status. The outcome measure was evaluated based on data from in-study observation period. In-study observation period is defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: Baseline (week 0), end of treatment (week 52)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 362 | 362
Scores on a scale | 2.0 [0.00 to 4.00] | 1.0 [-1.00 to 4.00]
Statistical Analysis 1: Comparison: Semaglutide vs Placebo; Test type: Superiority; p = 0.0108, Wilcoxon (Mann-Whitney); The Hodges-Lehmann estimate = 1.00, 95% CI 2-sided [0.478 to 1.518]

4. Secondary Outcome: Change in Pain-free Walking Distance on a Constant Load Treadmill Test
Description: Change in pain-free walking distance on a constant load treadmill test is presented. The constant-load treadmill test with fixed speed (3.2 km/h, 2 mph) and fixed inclination (12%) is a standardised method for functional assessment of patients with peripheral artery disease. Participants are instructed to when pain starts in either leg and to continue on the treadmill without stopping at this stage. The distance walked is noted as the pain-free walking distance. The outcome measure was evaluated based on data from in-study observation period. In-study observation period is defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: Baseline (week 0), end of treatment (week 52)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Ratio of pain-free walking distance
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 338 | 344
Ratio of pain-free walking distance | 1.21 [0.92 to 1.52] | 1.10 [0.86 to 1.44]
Statistical Analysis 1: Comparison: Semaglutide vs Placebo; Test type: Superiority; p = 0.0046, Wilcoxon (Mann-Whitney); The Hodges-Lehmann Estimate = 1.11, 95% CI 2-sided [1.033 to 1.197]

5. Secondary Outcome: Follow-up Change in Pain-free Walking Distance on a Constant Load Treadmill Test
Description: Change in pain-free walking distance on a constant load treadmill test is presented. The constant-load treadmill test with fixed speed (3.2 km/h, 2 mph) and fixed inclination (12%) is a standardised method for functional assessment of patients with peripheral artery disease. Participants are instructed to when pain starts in either leg and to continue on the treadmill without stop-ping at this stage. The distance walked is noted as the pain-free walking distance. The outcome measure was evaluated based on data from in-study observation period. In-study observation period is defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: Baseline (week 0), end of follow-up (week 57)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Ratio of pain-free walking distance
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 329 | 333
Ratio of pain-free walking distance | 1.18 [0.92 to 1.59] | 1.10 [0.83 to 1.48]

6. Secondary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change in HbA1c from baseline to week 52 in percentage-point is presented. The outcome measure is evaluated based on the on treatment without rescue treatment observation period. This period includes assessments and events for the time period where participants were exposed to trial product and before rescue treatment (medication or revascularisation procedure).
Time Frame: Baseline (week 0), end of treatment (week 52)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage-point of HbA1c
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 304 | 311
Percentage-point of HbA1c | -0.8 (1.1) | 0.2 (1.1)

7. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline to week 52 in kilogram (kg) is presented. The outcome measure is evaluated based on the on-treatment without rescue treatment observation period. This period includes assessments and events for the time period where participants were exposed to trial product and before rescue treatment (medication or revascularisation procedure).
Time Frame: Baseline (week 0), end of treatment (week 52)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 310 | 318
Kilogram (kg) | -5.2 (4.8) | -1.2 (4.2)

8. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change in systolic blood pressure from baseline to week 52 is presented.The outcome measure is evaluated based on the on treatment without rescue treatment observation period. This period includes assessments and events for the time period where participants were exposed to trial product and before rescue treatment (medication or revascularisation procedure).
Time Frame: Baseline (week 0), end of treatment (week 52)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimetre of mercury (mmHg)
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 310 | 319
Millimetre of mercury (mmHg) | -4 (15) | -1 (18)

9. Secondary Outcome: Change in Total Cholesterol
Description: Change in total cholesterol from baseline to week 52 is presented as ratio to baseline. The outcome measure is evaluated based on the on-treatment without rescue treatment observation period. This period includes assessments and events for the time period where participants were exposed to trial product and before rescue treatment (medication or revascularisation procedure).
Time Frame: Baseline (week 0), end of treatment (week 52)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 305 | 312
Ratio of total cholesterol | 0.96 (20.18) | 1.00 (19.88)

10. Secondary Outcome: Change in Low-density Lipoprotein (LDL)-Cholesterol
Description: Change in LDL-cholesterol from baseline to week 52 is presented as ratio to baseline. The outcome measure is evaluated based on the on-treatment without rescue treatment observation period. This period includes assessments and events for the time period where participants were exposed to trial product and before rescue treatment (medication or revascularisation procedure).
Time Frame: Baseline (week 0), end of treatment (week 52)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 294 | 296
Ratio of LDL | 0.99 (38.37) | 1.03 (42.27)

11. Secondary Outcome: Change in High Density Lipoprotein (HDL)-Cholesterol
Description: Change in HDL-cholesterol from baseline to week 52 is presented as ratio to baseline. The outcome measure is evaluated based on the on-treatment without rescue treatment observation period. This period includes assessments and events for the time period where participants were exposed to trial product and before rescue treatment (medication or revascularisation procedure).
Time Frame: Baseline (week 0), end of treatment (week 52)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 294 | 295
Ratio of HDL | 1.04 (15.95) | 0.99 (13.91)

12. Secondary Outcome: Change in Triglycerides
Description: Change in Triglycerides from baseline to week 52 is presented as ratio to baseline. The outcome measure is evaluated based on the on-treatment without rescue treatment observation period. This period includes assessments and events for the time period where participants were exposed to trial product and before rescue treatment (medication or revascularisation procedure).
Time Frame: Baseline (week 0), end of treatment (week 52)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 305 | 310
Ratio of triglycerides | 0.80 (45.95) | 0.95 (41.73)

13. Secondary Outcome: Change in Ankle-Brachial Index (ABI)
Description: Change in ABI from baseline to week 52 is presented. ABI is calculated as a ratio of the higher ankle systolic pressure to the higher systolic pressure measured in both arms. ABI is measured at both left and right leg and the analysis endpoint is defined as the lower of the two indices. An ABI between 1.0 to 1.4 is considered the normal range. An ABI between 0.90 to 0.99 is considered borderline. An ABI less than 0.90 indicates peripheral artery disease (PAD). The outcome measure is evaluated based on the on-treatment without rescue treatment observation period. This period includes assessments and events for the time period where participants were exposed to trial product and before rescue treatment (medication or revascularisation procedure).
Time Frame: Screening (week -2), end of treatment (week 52)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of ABI
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 306 | 315
Ratio of ABI | 1.06 (34.0) | 1.02 (19.6)

14. Secondary Outcome: Change in Toe-Brachial Index (TBI)
Description: Change in TBI from baseline to week 52 is presented. TBI is calculated as a ratio of the toe systolic pressure to the higher systolic pressure measured in both arms. TBI is measured at both left and right leg and the analysis endpoint is defined as the lower of the two indices. A TBI range of above or equal to 0.7 is considered normal, whereas a TBI less than 0.7 is considered abnormal. The outcome measure is evaluated based on the on-treatment without rescue treatment observation period. This period includes assessments and events for the time period where participants were exposed to trial product and before rescue treatment (medication or revascularisation procedure).
Time Frame: Screening (week -2), end of treatment (week 52)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of TBI
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 297 | 301
Ratio of TBI | 1.07 (34.4) | 1.04 (37.3)

15. Secondary Outcome: Change in Walking Impairment Questionnaire (WIQ) Global Score
Description: Change in WIQ global score from baseline to week 52 is presented. WIQ consists of three domains, speed, distance, and stair climbing, consisting of in total 14 questions. Each response is weighted based on the difficulty of the task. Domain scores are determined by dividing the weighted answers by the maximum possible weighted score and multiplying by 100. Global score is calculated as the mean of the three domain scores (ranged from 0% to 100%). A global score of 0% represents inabil-ity to perform any of the tasks and 100% represents no difficulty with any of the tasks. Higher scores indicate better walking ability and less impairment. The outcome measure is evaluated based on the on-treatment without rescue treatment observation period. This period includes assessments and events for the time period where participants were exposed to trial product and before rescue treatment (medication or revascularisation procedure).
Time Frame: Baseline (week 0), end of treatment (week 52)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: %-point scores on a scale
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 312 | 321
%-point scores on a scale | 9.48 (18.63) | 6.51 (20.53)

16. Secondary Outcome: Change in Short Form 36 (SF-36) Physical Functioning Domain
Description: Change in SF-36 physical functioning domain from baseline to week 52 is presented. SF-36 is a 36-item patient-reported survey of patient health that measures the participant's overall health-related quality of life (HRQoL). SF-36v2 (acute version) questionnaire measured 8 domains of functional health and well-being as well as 2 component summary scores (physical component summary and mental component summary). The 0-100 scale scores from the SF-36 were converted to norm-based scores (Range: 19.03 to 57.60) to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. A positive change score indicates an improvement in participant health stats. The outcome measure is evaluated based on the on-treatment without rescue treatment observation period. This period includes assessments and events for the time period where participants were exposed to trial product and before rescue treatment (medication or revascularisation procedure).
Time Frame: Baseline (week 0), end of treatment (week 52)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 311 | 320
Scores on a scale | 2.98 (7.32) | 1.52 (7.17)

ADVERSE EVENTS:
Time Frame: Until week 57
Description: All presented adverse events are treatment emergent adverse events (TEAEs). A Treatment Emergent Adverse Event (TEAE) is defined as an AE with onset in the on-treatment observation period.
Arm/Group | Semaglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 4/396 | 9/395
Serious Adverse Events (participants affected / at risk) | 74/396 | 78/395
Other Adverse Events (participants affected / at risk) | 47/396 | 24/395
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide (N=396) | Placebo (N=395)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Abdominal symptom (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Accelerated hypertension (Vascular disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 3 (5) | 5 (5)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 2 (2)
Angina unstable (Cardiac disorders) | 3 (3) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain abscess (Infections and infestations) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 2 (3) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 2 (3) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 2 (3) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Carotid artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 2 (3)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Cerebral infarction (Nervous system disorders) | 3 (3) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 4 (5) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 3 (3) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 3 (3) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
IIIrd nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Lacunar stroke (Nervous system disorders) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Optic nerve disorder (Eye disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 4 (4) | 5 (7)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 3 (3)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 5 (5)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rotavirus infection (Infections and infestations) | 1 (1) | 0 (0)
Scrotal ulcer (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Stomach mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tissue discolouration (General disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide (N=396) | Placebo (N=395)
COVID-19 (Infections and infestations) | 30 (32) | 21 (21)
Nausea (Gastrointestinal disorders) | 22 (26) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT04560998/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT04560998/SAP_001.pdf